CLINICAL TRIAL: NCT06000618
Title: Effects of Intrapulmonary Percussive Ventilator on Respiratory Function: an Experiment in Healthy Volunteers
Brief Title: Effects of Intrapulmonary Percussive Ventilator on Respiratory Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Sheng Wang MD PhD, MD PhD, Shanghai 10th People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STPH-ICU-006
Record Dates: First submitted 2023-07-20; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Airway Clearance Impairment
Keywords: Intrapulmonary percussive; Healthy volunteer; pulmonary function; Electrical Impedance Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): The experimental group will undergo intrapulmonary percussive therapy
  Interventions: Device: Intrapulmonary Percussive ventilator

INTERVENTIONS:
Device: Intrapulmonary Percussive ventilator — The volunteers will undergo three minutes low frequency and high frequency intrapulmonary percussive treatments.
  Other Names: MateNeb

SUMMARY:
The goal of this clinical trial is to prove the benefit of intrapulmonary percussive ventilator in healthy volunteers. The main questions are:

* How can intrapulmonary percussive improve lung function？
* What is the subjective feeling through intrapulmonary percussive?

Participants will be undergoing treatment of intrapulmonary percussive. Then they will be assessed for lung function and EIT before and after intrapulmonary percussive.

ELIGIBILITY:
Inclusion Criteria:

* No respiratory system, heart disease
* Well cooperate with the MateNeb

Exclusion Criteria:

* No respiratory illness such as influenza, pneumonia, asthma, bronchitis within the last month
* Couldn't finish three times pulmonary function test

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Pulmonary function test | through study completion, an average one hour
  This test can assess the volunteer's lung ventilation and diffusion function.For example the max vital capacity (VCMAX),Forced vital capacity(FVC),Forced expiratory volume in one second(FEV1),functional residual capacity(FRC-SB),diffusion capacity of lung for carbon monoxide(DLCO) and so on.
Electrical Impedance Tomography of Pulmonary(EIT) | through study completion, an average one hour
  EIT is a relatively advanced non-invasive monitoring technique for the lung function. This technology uses a strap attached to the chest to monitor electrical at 16 locations. The Ventilation in each area resistance of the lung is quantified according to the electrical resistance

SECONDARY OUTCOMES:
The safety and comfort | The treatment was scored once after the participants completed both low and high frequency intrapulmonary percussive.Up to one week.
  Whether the technique has adverse reactions. How do the volunteers feel? We used a scale of 1 to 4 to show how the volunteers felt. 1 is the worst feeling. The volunteers were no longer willing to undergo the treatment. 4 means the volunteers felt better and breathed easier after the treatment. Be willing to undergo endoairway shock therapy again.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng Wang, PHD, Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hassan A, Milross M, Lai W, Shetty D, Alison J, Huang S. Feasibility and safety of intrapulmonary percussive ventilation in spontaneously breathing, non-ventilated patients in critical care: A retrospective pilot study. J Intensive Care Soc. 2021 May;22(2):111-119. doi: 10.1177/1751143720909704. Epub 2020 Mar 12. PMID 34025750
- [Result] Nyland BA, Spilman SK, Halub ME, Lamb KD, Jackson JA, Oetting TW, Sahr SM. A Preventative Respiratory Protocol to Identify Trauma Subjects at Risk for Respiratory Compromise on a General In-Patient Ward. Respir Care. 2016 Dec;61(12):1580-1587. doi: 10.4187/respcare.04729. Epub 2016 Nov 8. PMID 27827332